CLINICAL TRIAL: NCT07179588
Title: Dietary Intervention to Reduce Pain in Spinal Cord Injury
Brief Title: Nutrition and Pain Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Academy of Spinal Cord Injury Professionals, Inc. (Unknown)
Responsible Party: Principal Investigator, Elizabeth Felix, Research Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250188
Record Dates: First submitted 2025-09-16; First posted 2025-09-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: SCI - Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Group (Experimental): Participants will be in this group for up to 4 months.
  Interventions: Behavioral: Nutrition Education Program; Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Nutrition Education Program — The participants will attend a monthly nutrition education session for 4 months (total 4 sessions). The sessions will be available in person and over teleconference platforms (i.e., Zoom). Each session will be up to 1-hour, which will include nutrition guidelines to manage diet quality.
Behavioral: Nutrition Counseling — Participant will meet with a registered dietitian for one-on-one diet consults once a month for 4 months. These sessions can be in-person or via Zoom. Each session will be up to 1 hour, and will be done to assess if the nutrition guidelines taught during the education sessions are being implemented.

SUMMARY:
The purpose of this research is to assess the effectiveness of a nutrition intervention on diet quality in managing pain in individuals with spinal cord injury (SCI).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 y)
* With SCI (motor complete or incomplete American Spinal Injury Association Impairment Scale (AIS) A-D, paraplegia or ventilator-independent tetraplegia)
* Have chronic pain

Exclusion Criteria:

* Adults unable to consent Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women (self-report)
* Prisoners
* Those not meeting inclusion criteria will be excluded (e.g., no pain).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain rating as measured by the Numerical Rating Scale | Baseline, 4-months (after intervention)
  The primary pain outcome will be measured using a 0 to 10 numerical rating scale (NRS) of average pain intensity during the past week, with higher scores indicating higher pain intensity.
Change in neuropathic pain severity as measured by the Neuropathic Pain Symptom Inventory | Baseline, 4-months (after intervention)
  Neuropathic pain severity outcome will be measured using the Neuropathic Pain Symptom Inventory (NPSI; 0-100) with higher scores indicating greater pain levels. This neuropathic pain rating will be captured at baseline and after the intervention period (4 months).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Felix, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No